CLINICAL TRIAL: NCT02945371
Title: Tailored Inhibitory Control Training to Reverse EA-linked Deficits in Mid-life
Acronym: REV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPCS20613
Record Dates: First submitted 2016-03-25; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Smoking; Alcohol Drinking; Prescription Drug Abuse; Substance-Related Disorders; Oral Intake Reduced
MeSH Terms: conditions — Smoking; Alcohol Drinking; Substance-Related Disorders | interventions — 26S proteasome non-ATPase regulatory subunit 13; JPT1 protein, human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IC Training (Experimental): The experimental arm (ARM1) is a "person-centered inhibitory control" training intervention, or PeCIC.
  Between the baseline and endpoint sessions, participants come to our lab 12 times to participate in the training sessions. Each participant is randomly assigned to either the PeCIC training or an active control training. The training sessions will take place approx. every other day for 24 days.
  Beginning 2-3 days after the baseline session, the experimental group (will come to our behavioral testing lab to receive the PeCIC training. At 11 sessions spaced one every other day, participants will complete one 8-min run of a modified stop-signal task. The cue on each trial (preceding the "go" signal arrow) will be an image of a personalized risk-cue (PRC) or a neural image.
  Interventions: Behavioral: Person-centered inhibitory control training
- Control Training (Active Comparator): Participants in the active control group (ARM2) of the PeCIC intervention will come to the behavioral testing laboratory to complete an 8-min control task every other day for 12 sessions. This control task is identical to the PeCIC except the auditory stop cues are omitted. All other procedures, settings, and schedules are identical to those in the experimental group. The only difference between the groups is that the active control does not practice IC.
  Interventions: Behavioral: Active behavioral response training

INTERVENTIONS:
Behavioral: Person-centered inhibitory control training — A brief, computer-based, multisession training aimed at increasing the connection between environmental risk cues (e.g., cigarettes) and engagement of the brain network for inhibitory control.
  Other Names: PeCIC, ARM1
  Arms: IC Training
Behavioral: Active behavioral response training — A brief computer-based, multisession training aimed at training behavioral responses to personalized environmental risk cues (e.g., cigarettes) that does not engage the inhibitory control network of the brain.
  Other Names: Active control, ARM2
  Arms: Control Training

SUMMARY:
Insufficient inhibitory control is one pathway through which early adversity is related to a range of problems including excessive alcohol use, tobacco use, and unhealthy eating. The proposed research leverages a neurally informed model of inhibitory control and how it can be improved to test the efficacy of a person-centered inhibitory control intervention in a sample of mid-life individuals with early adversity. The knowledge obtained by this study could be scaled into a flexible, low-cost, and wide-ranging intervention to remediate some of the effects of early adversity on inhibitory control and thus a number of prevalent health risking behaviors.

DETAILED DESCRIPTION:
Early adversity (EA) in humans is a major contributing factor to a range of deleterious physical and mental health outcomes extending through adulthood such as depression and anxiety, obesity and heart disease, and premature death. In addition to detracting significantly from individual well being and quality of life, these conditions also consume considerable resources from federal, state, and community organizations. The mechanisms through which EA exerts its effects on these outcomes are increasingly well understood, and include neurocognitive pathways related to executive function. An intervention that can successfully target, engage with, and alter the functioning of one or more of these mechanisms would be a promising way of mitigating the impact of EA on deleterious outcomes later in life. The proposed research focuses on one such pathway-deficits in inhibitory control (IC)-and tests the feasibility and efficacy of an intervention to increase functioning in that pathway in a sample of individuals who experienced EA. The intervention is grounded in a neurally informed model of change that specifies deficits in IC as an underlying causal factor common to several health-risking behaviors (HRBs). These IC deficits emerge during development as a result of a range of EA, and, critically, can be remediated in mid-life through targeted intervention. Research from our laboratory has validated an intervention that can increase IC performance and alter its underlying neural systems in young adults (Berkman, Kahn, & Merchant, 2014). The next step in this program of research, proposed here, is to test the efficacy of that intervention in a sample of mid-life individuals who have experienced EA and the extent to which our intervention generalizes to HRBs that are prevalent in that sample. The first Aim is to test whether the intervention alters the IC system in tasks both similar to and dissimilar from the training task in terms of both behavioral performance and neural functioning. The second Aim is to test whether alterations in the functioning of the underlying neural systems mediate the effect of the intervention on performance and disinhibition-related HRBs. The two Aims will be accomplished within the context of a single randomized controlled trial (RCT) with two arms (IC training vs. active control) and pre-post measurements of IC performance, IC neural systems, and HRBs. All participants (N = 110) come to the lab for an initial assessment of behavioral / neural measures of IC and HRBs, among other measures. Then, participants are randomly assigned to receive a Person-Centered Inhibitory Control (PeCIC) training or active control training, every other day for 3-4 weeks. The PeCIC systematically pairs IC engagement with alcohol, tobacco, and/or energy-dense food cues, depending on each participant's reports of disinhibited behavior in those domains. The active control task uses personalized cues and response time tasks but does not involve IC. Finally, participants return to the laboratory for an endpoint assessment where all baseline measures are repeated. The two Aims will be robustly tested in a series of analyses comparing the behavioral and neural change from pre- to postintervention between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-55
* Experience of early adversity (EA) before age 18 (EA is be defined as a score of 4 or higher on the Adverse Childhood Experiences (ACEs) questionnaire [Felitti, Anda, Nordenberg, Williamson, Spitz, Edwards, et al., 1998])
* IC difficulties such as disinhibited alcohol use, tobacco use, or food intake during adulthood. IC difficulties will be self-reported based on questions from the self-control questionnaire (Tangney, Baumeister, & Boone, 2004) modified to be specific to alcohol, tobacco, and energy-dense food intake (e.g., "I am self-indulgent with unhealthy food at times", "I refuse alcohol when offered") using a 4-point Likert-style scale.

Exclusion Criteria:

* Individuals over age 55 will be excluded because of established functional and structural neural changes that begin to escalate at that time (Good, Johnsrude, Ashburner, Henson, Friston, & Frackowiak, 2001; Grady, Springer, Hongwanishkul, McIntosh, & Winocur, 2006)
* Given the high rates of morbidity for such disorders among people with high EA, we will not exclude based on past diagnoses for any of those disorders or based on current drug and alcohol use. However, we will exclude individuals who do not pass a urine toxicology screen during either of the functional magnetic resonance imaging (fMRI) sessions to ensure that the neuroimaging data are as homogeneous and reliable as possible.
* Participants who cannot undergo an MRI scan will be excluded; contraindications include metal implants (e.g., braces, pins) or metal fragments, pacemakers or other electronic medical implants, claustrophobia, pregnancy, and weight greater than 550 lbs.

Beyond these criteria, participants will be recruited without exclusions based on gender, race, or ethnicity, so our sample will reflect the diversity in the local population (Lane County, Oregon) with regard to gender, race, and ethnicity.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Inhibitory control performance, Task 1 | 1 month
  Performance on a standard inhibitory control task (Stop-Signal) with personal risk cues
Inhibitory control performance, Task 2 | 1 month
  Performance on a standard inhibitory control task (Go/No-Go) with personal risk cues
Inhibitory control neural activity | 1 month
  Early ("proactive") engagement of the inferior frontal gyrus and dorsal anterior cingulate cortex during the inhibitory control tasks

SECONDARY OUTCOMES:
Far transfer to a task related to inhibitory control, Behavioral marker | 1 month
  Performance on a standard risky-behavior task (Balloon Analogue Risk task)
Far transfer to a task related to inhibitory control, Neural marker | 1 month
  Neural activity during a standard risky-behavior task (Balloon Analogue Risk task)
Health-risking behavior | 1 month, 3 months
  Standard self-report questions regarding health-risking behavior related to inhibitory control (e.g., cigarette smoking, excessive alcohol intake, illicit drug use and prescription drug misuse, and excessive energy intake)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot T Berkman, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Social and Affective Neuroscience Laboratory, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher PA, Berkman ET. Designing Interventions Informed by Scientific Knowledge About Effects of Early Adversity: A Translational Neuroscience Agenda for Next Generation Addictions Research. Curr Addict Rep. 2015 Dec 1;2(4):347-353. doi: 10.1007/s40429-015-0071-x. Epub 2015 Sep 28. PMID 26985399
- [Background] Berkman ET, Lukinova E, Menshikov I, Myagkov M. Sociality as a natural mechanism of public goods provision. PLoS One. 2015 Mar 19;10(3):e0119685. doi: 10.1371/journal.pone.0119685. eCollection 2015. PMID 25790099
- [Background] Giuliani NR, Tomiyama AJ, Mann T, Berkman ET. Prediction of daily food intake as a function of measurement modality and restriction status. Psychosom Med. 2015 Jun;77(5):583-90. doi: 10.1097/PSY.0000000000000187. PMID 25984820
- See also: Social and Affective Neuroscience (SAN) Laboratory website — http://sanlab.uoregon.edu
- See also: Study recruitment website — http://sanlab.uoregon.edu/participate/